CLINICAL TRIAL: NCT03669588
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase 3 Trial to Evaluate the Efficacy, Safety and Tolerability of ARGX-113 in Patients With Myasthenia Gravis Having Generalized Muscle Weakness
Brief Title: An Efficacy and Safety Study of ARGX-113 in Patients With Myasthenia Gravis Who Have Generalized Muscle Weakness
Acronym: ADAPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-1704; 2018-002132-25 (EudraCT Number)
Expanded Access: NCT04777734 (Approved for marketing)
Record Dates: First submitted 2018-09-06; First posted 2018-09-13 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-03

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — efgartigimod alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARGX-113 (Experimental)
  Interventions: Biological: ARGX-113
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ARGX-113 — Intravenous administration of ARGX-113
  Other Names: efgartigimod
  Arms: ARGX-113
Biological: Placebo — Intravenous administration of placebo
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo controlled, multicenter Phase 3 trial to evaluate the efficacy, safety, tolerability, quality of life and impact on normal daily activities of ARGX-113 in patients with gMG.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the ability to understand the requirements of the trial, provide written informed consent, and comply with the trial protocol procedures.
2. Male or female patients aged ≥ 18 years.
3. Diagnosis of MG with generalized muscle weakness meeting the clinical criteria for diagnosis of MG as defined by the Myasthenia Gravis Foundation of America (MGFA) class II, III, IVa and IVb.

Other, more specific inclusion criteria are defined in the protocol

Exclusion Criteria:

1. Pregnant and lactating women, and those intending to become pregnant during the trial or within 90 days after the last dosing.
2. Male patients who are sexually active and do not intend to use effective methods of contraception during the trial or within 90 days after the last dosing or male patients who plan to donate sperm during the trial or within 90 days after the last dosing.
3. MGFA Class I and V patients.
4. Patients with worsening muscle weakness secondary to concurrent infections or medications.
5. Patients with known seropositivity or who test positive for an active viral infection at Screening with:

   * Hepatitis B Virus (HBV) (except patients who are seropositive because of HBV vaccination)
   * Hepatitis C Virus (HCV)
   * Human Immunodeficiency Virus (HIV)

Other, more specific exclusion criteria are further defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Guglietta, MD, Study Director — argenx
Locations (66):
- United States (25):
  - Investigator Site 29, Phoenix, Arizona
  - Investigator Site 66, Carlsbad, California
  - Investigator Site 5, Los Angeles, California
  - Investigator Site 49, Los Angeles, California
  - Investigator Site 18, Orange, California
  - Investigator Site 40, Palo Alto, California
  - Investigator Site 59, San Francisco, California
  - Investigator Site 58, Aurora, Colorado
  - Investigator Site 34, Jacksonville, Florida
  - Investigator Site 4, Tampa, Florida
  - Investigator Site 30, Springfield, Illinois
  - Investigator Site 25, Iowa City, Iowa
  - Investigator Site 21, Kansas City, Kansas
  - Investigator Site 27, Boston, Massachusetts
  - Investigator Site 48, Detroit, Michigan
  - Investigator Site 53, Buffalo, New York
  - Investigator Site 3, Chapel Hill, North Carolina
  - Investigator Site 20, Cleveland, Ohio
  - Investigator Site 9, Portland, Oregon
  - Investigator Site 17, Charleston, South Carolina
  - Investigator Site, Cordova, Tennessee
  - Investigator Site 44, Houston, Texas
  - Investigator Site 6, San Antonio, Texas
  - Investigator Site 2, Charlottesville, Virginia
  - Investigator Site 16, Seattle, Washington
- Belgium (2):
  - Investigator Site 11, Edegem
  - Investigator Site 8, Ghent
- Canada (3):
  - Investigator Site 38, Edmonton, Alberta
  - Investigator Site 24, Toronto, Ontario
  - Investigator Site 22, Montreal, Quebec
- Czechia (3):
  - Investigator Site 32, Brno
  - Investigator Site 35, Ostrava-Poruba
  - Investigator Site 51, Prague
- Denmark (2):
  - Investigator Site 36, Aarhus
  - Investigator Site 15, Copenhagen
- France (2):
  - Investigator Site 13, Bordeaux
  - Investigator Site 52, Marseille
- Georgia (3):
  - Investigator Site 46, Tbilisi
  - Investigator Site 45, Tbilisi
  - Investigator Site 47, Tbilisi
- Investigator Site 33, Berlin, Germany
- Hungary (2):
  - Investigator Site 55, Budapest
  - Investigator Site 54, Szeged
- Italy (2):
  - Investigator Site 10, Milan
  - Investigator Site 12, Napoli
- Japan (9):
  - Investigator Site 42, Chiba, Chiba
  - Investigator Site 26, Sapporo, Hokkaido
  - Investigator Site 19, Hanamaki, Iwate
  - Investigator Site 43, Sendai, Miyagi
  - Investigator Site 28, Ōsaka-sayama, Osaka
  - Investigator Site 50, Suita, Osaka
  - Investigator Site 31, Meguro City, Tokyo
  - Investigator Site 41, Minato-Ku, Tokyo
  - Investigator Site 39, Shinjuku-Ku, Tokyo
- Investigator Site 37, Leiden, Netherlands
- Poland (4):
  - Investigator Site 7, Gdansk
  - Investigator Site 57, Katowice
  - Investigator Site 14, Krakow
  - Investigator Site 23, Warsaw
- Russia (4):
  - Investigator Site 64, Krasnoyarsk
  - Investigator Site 62, Nizhny Novgorod
  - Investigator Site 65, Novosibirsk
  - Investigator Site 60, Samara
- Investigator Site 61, Belgrade, Serbia
- United Kingdom (2):
  - Investigator Site 63, Edgbaston
  - Investigator Site 56, Liverpool

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoffmann S, Zhao S, Callewaert F, Schoppe S, Rozsa C, Spillane J. Post Hoc, Sex-Specific Subgroup Analysis of Efgartigimod in Patients With Generalized Myasthenia Gravis From the ADAPT Trial: A Sex and Gender Equity in Research (SAGER) Guidelines Approach. Muscle Nerve. 2026 Jan 10. doi: 10.1002/mus.70135. Online ahead of print. PMID 41517964
- [Derived] Janssen MF, Dewilde S, Wolfe GI, Muppidi S, Phillips G. Psychometric properties of MG-ADL items and MG-ADL score: An assessment of distributional characteristics, validity and factor structure in two large datasets. J Neurol Sci. 2024 Aug 15;463:123135. doi: 10.1016/j.jns.2024.123135. Epub 2024 Jul 22. PMID 39068745
- [Derived] Howard JF Jr, Bril V, Vu T, Karam C, Peric S, Margania T, Murai H, Bilinska M, Shakarishvili R, Smilowski M, Guglietta A, Ulrichts P, Vangeneugden T, Utsugisawa K, Verschuuren J, Mantegazza R; ADAPT Investigator Study Group. Safety, efficacy, and tolerability of efgartigimod in patients with generalised myasthenia gravis (ADAPT): a multicentre, randomised, placebo-controlled, phase 3 trial. Lancet Neurol. 2021 Jul;20(7):526-536. doi: 10.1016/S1474-4422(21)00159-9. PMID 34146511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in generalized myasthenia gravis (gMG) patients at 56 sites worldwide. Patients were randomized 1:1 within each stratum (Japanese/non-Japanese, acetylcholine receptor-antibody [AChR-Ab] status and standard of care [SoC; ie, concomitant gMG treatment]) to receive ARGX-113 intravenous (IV) 10 milligrams/kilogram (mg/kg) or placebo, in addition to SoC. Patients completing the study were eligible to roll over into a follow-up study ARGX-113-1705.
Pre-assignment Details: Total study duration was up to 28 weeks, including a 2-week screening period, an initial 8-week treatment cycle (TC) and intertreatment cycle (ITC) of variable length depending on the patient. Patients had to be on a stable dose of SoC and not have received immunoglobulins by IV, subcutaneous or intramuscular route, or plasma exchange, < 1 month prior to screening. The study included both AChR-Ab seropositive and seronegative patients; AChR-Ab detection in serum was performed during screening.
Groups:
- ARGX-113: Patients received ARGX-113 IV 10 mg/kg administered as a 1-hour infusion every 7 days for 4 infusions (Days 1, 8, 15, and 22) in each cycle.
  Each 8-week TC comprised a 3-week treatment period and a 5-week follow-up period. At the end of each TC, patients entered the ITC period consisting of visits every 2 weeks. At each ITC visit, retreatment criteria were evaluated to determine if the patient was eligible to enter the next cycle for retreatment, based on clinical response as measured by the Myasthenia Gravis Activities of Daily Living (MG-ADL) scale.
- Placebo: Patients received matching placebo administered as a 1-hour infusion every 7 days for 4 infusions (Days 1, 8, 15, and 22) in each cycle.
  Each 8-week TC comprised a 3-week treatment period and a 5-week follow-up period. At the end of each TC, patients entered the ITC period consisting of visits every 2 weeks. At each ITC visit, retreatment criteria were evaluated to determine if the patient was eligible to enter the next cycle for retreatment, based on clinical response as measured by the MG-ADL scale.
Period: Overall Study
Arm/Group | ARGX-113 | Placebo
Started | 84 | 83
Completed | 80 | 76
Not Completed | 4 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Sponsor Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Rescue Therapy Needed | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients in the randomized population who received at least a partial dose of investigational medicinal product (IMP) were included in the baseline analysis.
Groups:
- ARGX-113: Patients received ARGX-113 IV 10 mg/kg administered as a 1-hour infusion every 7 days for 4 infusions (Days 1, 8, 15, and 22) in each cycle.
- Placebo: Patients received matching placebo administered as a 1-hour infusion every 7 days for 4 infusions (Days 1, 8, 15, and 22) in each cycle.
- Total: Total of all reporting groups
Arm/Group | ARGX-113 | Placebo | Total
Number analyzed (Participants) | 84 | 83 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (14.41) | 48.2 (14.97) | 47.0 (14.69)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 73 | 69 | 142
  >= 65 years | 11 | 14 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 55 | 118
  Male | 21 | 28 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 9 | 7 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 69 | 72 | 141
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 8 | 7 | 15
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 69 | 73 | 142
  Not Reported | 0 | 1 | 1
Concomitant gMG treatment [Count of Participants; unit: Participants]
  Nonsteroidal Immunosuppressive Drugs (NSIDs) | 51 | 51 | 102
  No NSIDs | 33 | 32 | 65
AChR-Ab status [Count of Participants; unit: Participants]
  Positive | 65 | 64 | 129
  Negative | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of MG-ADL Responders During Cycle 1 (C1); Analyzed in the AChR-Ab Seropositive Population
Description: The MG-ADL is an 8-item patient-reported scale to assess MG symptoms and their effects on daily activities. The scale comprises 2 items on daily life activities and 6 items on symptoms. The MG-ADL total score range is 0-24, with higher scores indicative of greater disease severity. A patient was considered an MG-ADL responder during C1 if there was a reduction of ≥2 points on the MG-ADL total score (compared to baseline of C1 [C1B]) for ≥4 consecutive weeks with the first reduction occurring no later than 1 week after the last infusion of IMP in C1.
Time Frame: Baseline up to Day 63 (end of TC1)
Population: Analysis was performed in the AChR-Ab seropositive population using the modified intention-to-treat (mITT) analysis set which included all randomized patients with a value for the MG-ADL total score at baseline and at least 1 postbaseline timepoint.
Measure: Number; unit: percentage of patients
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 65 | 64
percentage of patients | 67.7 | 29.7
Statistical Analysis 1: Comparison: ARGX-113 vs Placebo; Analysis with a 2-sided exact test (using logistic regression) at the 2-sided 5% significance level in the AChR-Ab seropositive population, stratified by Japanese versus (vs) non-Japanese and NSID vs no NSID as concomitant gMG treatment, with cycle baseline MG-ADL total score as covariate. The treatment effect was presented as the odds ratio. An odds ratio of more than 1 represents a higher response rate for ARGX-113 compared to placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.951, 95% CI 2-sided [2.213 to 11.528]

2. Secondary Outcome: Percentage of Quantitative Myasthenia Gravis (QMG) Responders During C1; Analyzed in the AChR-Ab Seropositive Population
Description: The QMG scale quantifies disease severity based on impairments of body functions and structures as defined by the International Classification of Disability and Health. The QMG scale consists of 13 items that measure endurance or fatigability, and accounts for fluctuations in disease state. The QMG total score range is 0-39, with higher scores indicative of greater disease severity. A patient was considered a QMG responder during C1 if there was a reduction of ≥3-points on the QMG total score (compared to C1B) for ≥4 consecutive weeks with the first reduction occurring no later than 1 week after the last infusion of IMP in C1.
Time Frame: Baseline up to Day 63 (end of TC1)
Population: Analysis was performed in the AChR-Ab seropositive population using the mITT analysis set which included all randomized patients with a value for the MG-ADL total score at baseline and at least 1 postbaseline timepoint.
Measure: Number; unit: percentage of patients
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 65 | 64
percentage of patients | 63.1 | 14.1
Statistical Analysis 1: Comparison: ARGX-113 vs Placebo; Analysis with a 2-sided exact test (using logistic regression) at the 2-sided 5% significance level in the AChR-Ab seropositive population, stratified by Japanese vs non-Japanese and NSID vs no NSID as concomitant gMG treatment, with cycle baseline QMG total score as covariate. The treatment effect was presented as the odds ratio. An odds ratio of more than 1 represents a higher response rate for ARGX-113 compared to placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 10.842, 95% CI 2-sided [4.179 to 31.200]

3. Secondary Outcome: Percentage of MG-ADL Responders During C1; Analyzed in the Overall Population
Description: The percentage of MG-ADL responders during C1 in the overall population is reported for this secondary end point; percentage of MG-ADL responders during C1 in the AChR-Ab seropositive population is reported previously as a primary end point.
Time Frame: Baseline up to Day 63 (end of TC1)
Population: Analysis was performed in the overall population (including both AChR-Ab seropositive and seronegative patients) using the mITT analysis set which included all randomized patients with a value for the MG-ADL total score at baseline and at least 1 postbaseline timepoint.
Measure: Number; unit: percentage of patients
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 84 | 83
percentage of patients | 67.9 | 37.3
Statistical Analysis 1: Comparison: ARGX-113 vs Placebo; Analysis with a 2-sided exact test (using logistic regression) at the 2-sided 5% significance level in the overall population, stratified by AChR-Ab status (seropositive vs seronegative), Japanese vs non-Japanese and NSID vs no NSID as concomitant gMG treatment, with cycle baseline MG-ADL total score as covariate. The treatment effect was presented as the odds ratio. An odds ratio of more than 1 represents a higher response rate for ARGX-113 compared to placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.699, 95% CI 2-sided [1.854 to 7.578]

4. Secondary Outcome: Percentage of Time That Patients Had a Clinically Meaningful Improvement (CMI) in MG-ADL Total Score up to and Including Day 126; Analyzed in the AChR-Ab Seropositive Population
Description: An MG-ADL CMI was defined as a reduction of ≥2 points on the total MG-ADL score compared to study entry baseline (SEB).
Time Frame: Baseline up to Day 126
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 65 | 64
percentage of time | 48.714 (6.163) | 26.649 (6.316)
Statistical Analysis 1: Comparison: ARGX-113 vs Placebo; Analysis of covariance (ANCOVA) in the AChR-Ab seropositive population with treatment, baseline MG-ADL total score, Japanese vs non-Japanese, and NSID vs no NSID as concomitant gMG treatment as the covariates; Test type: Superiority; p = 0.0001, ANCOVA; Least square means difference = 22.065, 95% CI 2-sided [10.949 to 33.181], Standard Error of Mean 5.616

5. Secondary Outcome: Time From Week 4 to Qualify for Retreatment; Analyzed in the AChR-Ab Seropositive Population
Description: Time to qualify for retreatment was defined as time from the Week 4 assessment until the first visit with a <2-point reduction compared to SEB in the MG-ADL total score and MG-ADL total score ≥5 points with >50% of the total score attributable to nonocular symptoms.
Time Frame: Week 4 up to Day 182 (end of study [EoS])
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 65 | 64
days | 35.0 [29.0 to 43.0] | 8.0 [1.0 to 30.0]
Statistical Analysis 1: Comparison: ARGX-113 vs Placebo; Analysis was performed in the AChR-Ab seropositive population and the p-value was calculated using the log-rank test, stratified by Japanese vs non-Japanese and NSID vs no NSID as concomitant gMG treatment; Test type: Superiority; p = 0.2604, Log Rank

6. Secondary Outcome: Percentage of Early MG-ADL Responders During C1; Analyzed in the AChR-Ab Seropositive Population
Description: A patient was considered an early MG-ADL responder during C1 if there was a reduction of ≥2 points on the MG-ADL total score (compared to C1B) for ≥4 consecutive weeks with the first reduction occurring no later than Week 2 (ie, after 1 or maximum 2 infusions of IMP in C1).
Time Frame: Baseline up to Day 63 (end of TC1)
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 65 | 64
percentage of patients | 56.9 | 25.0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were monitored from first administration of IMP on Day 1 until the EoS (up to a maximum of approximately 182 days).
Description: The safety analysis set included patients in the randomized population who received at least a partial dose of IMP.
Arm/Group | ARGX-113 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/83
Serious Adverse Events (participants affected / at risk) | 4/84 | 7/83
Other Adverse Events (participants affected / at risk) | 49/84 | 48/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARGX-113 (N=84) | Placebo (N=83)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Therapeutic product ineffective (General disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 2 (2)
Myasthenia gravis crisis (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARGX-113 (N=84) | Placebo (N=83)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 9 (14)
Nausea (Gastrointestinal disorders) | 7 (7) | 9 (15)
Bronchitis (Infections and infestations) | 5 (6) | 2 (2)
Nasopharyngitis (Infections and infestations) | 10 (12) | 15 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (3)
Dizziness (Nervous system disorders) | 3 (5) | 5 (5)
Headache (Nervous system disorders) | 24 (40) | 23 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Hypertension (Vascular disorders) | 3 (4) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 4 (4)
Urinary tract infection (Infections and infestations) | 8 (9) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT03669588/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT03669588/SAP_001.pdf